CLINICAL TRIAL: NCT06499974
Title: Impact of Preoperative Anemia Severity and Classification on Perioperative Oxygen Supply-Demand Imbalance-Related Complications--A Prospective Observational Multi-center Cohort Study
Brief Title: POASAC Study (Preoperative Anemia Severity and Classification Study)
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: K3049
Record Dates: First submitted 2024-06-26; First posted 2024-07-15 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2024-12

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- IDA: patients with iron-deficiency anemia
- ACD/AI: patients with anemia of chronic disease/anemia of inflammation
- Combined anemia: patients with IDA and ACD/AI

SUMMARY:
The goal of this observational study focuses on the effect of different preoperative anemia status on perioperative complications in patients under moderate- to high-risk surgery. Different anemia types conclude iron-deficiency anemia(IDA), anemia of chronic disease/anemia of inflammation(ACD/AI), and combined anemia.The main question it aims to answer is whether there is a difference in the incidence of complication related to oxygen supply and demand imbalance in patients with IDA, ACD/AI or combined anemia.

Patients without preoperative anemia will be recruited as the control group for secondary outcome analysis, which is whether there is a difference in the incidence of complication related to oxygen supply and demand imbalance in patients with or without anemia.

DETAILED DESCRIPTION:
The investigators aim to screen patients according to including and excluding criteria. According to the hemoglobin level, if the patient is anemia, the investigators will offer some lab tests for serum iron, transferrin saturation, C-reactive protein to classify different anemia status. Besides, the investigators will include patients without anemia in a 2:1 ration of anemia to non-anemia. The perioperative assessment and follow-up are the same for all the included patients.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* scheduled for elective moderate- to high-risk surgery other than intracranial and cardiac surgery
* predicted surgery time longer than 1 hour and hospital stay longer than 24 hours
* understand and agree to participate

Exclusion Criteria:

* pregnant
* live at areas higher than 2,500 meters above sea level
* with hematological diseases other than anemia
* with severe comorbidities that might interfere outcome assessment, like uremia, dementia, and so on
* can't cooperate or communicate, or reject to sign informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are 18 years or older scheduled for moderate- or high-risk surgery will be included in our study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-08-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
postoperative complications related to oxygen supply and demand imbalance | before discharge or until seven days after surgery
  The occurrence of any of the following complications is considered a positive outcome, which include myocardial injury after non cardiac surgery(MINS), acute kidney injury(AKI), neurological damage such as stroke and delayed neurocognitive recovery(DNR)

SECONDARY OUTCOMES:
The incidence of post complications related to oxygen supply and demand imbalance in patients with or without anemia | before discharge or seven days after surgery
  The occurrence of any of the following complications is considered a positive outcome, which include myocardial injury after non cardiac surgery(MINS), acute kidney injury(AKI), neurological damage such as stroke and delayed neurocognitive recovery(DNR)
Postoperative functional disability | 1 month, 6 months and 1 year after surgery
  The World Health Organization Disability Assessment Schedule 2.0 (WHO DAS2.0) is used for disability assessment.
Cognitive function decline | 1 month, 6 months and 1 year after surgery
  The modified Telephone Interview for Cognitive Status(TICS-m) is used for cognitive function assessment.
RBC Transfusion rate | From date of surgery until discharge day, assessed up to 4 weeks
  The above information can be got according to the medical record
Length of hospital stay | From date of surgery until discharge day, assessed up to 4 weeks
  The above information can be got according to the medical record
Severe complication | before discharge, 1 month, 6 months and 1 year after surgery
  Evaluated according to Clavien-Dindo classification, level three to five are defined as severe complication.

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - Department of Anesthesiology, First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Beijing Longfu Hospital (Beijing Geriatric Hospital of Integrated Traditional Chinese and Western Medicine), Beijing, Beijing Municipality
  - Anesthesiology Department, Beijing NO.6 Hospital, Beijing, Beijing Municipality
  - BeiJing Hepingli Hospital, Beijing, Beijing Municipality
  - Beijing Puren Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Science and Education Department, Zhangzhou Municipal Hospital of Fujian Province, Zhangzhou, Fujian
  - Department of Anesthesiology, Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - Department of Anesthesiology, Chifeng Municipal Hospital, Chifeng, Inner Mongolia
  - Department of Anesthesiology, The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Inner Mongolia People's Hospital, Hohhot, Inner Mongolia